CLINICAL TRIAL: NCT01645722
Title: Enriched Autologous Fat Grafting for Treating Pain at Amputation Sites
Acronym: AMP-5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO11090215
Record Dates: First submitted 2012-03-21; First posted 2012-07-20 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Amputation Stumps; Pain
Keywords: Fat Grafts; Autogenous Fat Transfers (AFT); Wounded warriors; Amputation pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Procedure/Surgery: Enriched Fat grafting (Other): Enriched Fat grafting
  Interventions: Procedure: Procedure/Surgery: Enriched Fat grafting

INTERVENTIONS:
Procedure: Procedure/Surgery: Enriched Fat grafting — Fat grafting is a minimally invasive clinical procedure that has been widely used by plastic surgeons within reconstructive surgery for many years. Fat tissue to be used for grafting is harvested (usually from abdomen or thighs) in the operating room. The fat tissue is then sterilely centrifuged and allowed to decant before separating the fluid and oil layers from the fat tissue fraction. The aspirated fat is then injected into the amputation stump.In this study, we will concentrate the adipose stromal cells (ASCs) in the fat graft material to assess whether this modification will increase fat graft retention over time. The volume retention in areas treated with ASC concentrated fat grafts will be compared with regions treated with standard fat grafts in the same patient.
  Other Names: Fat Grafts; Autogenous Fat Transfers (AFT); Wounded warriors; Amputation site pain; Amputation pain

SUMMARY:
The objective of this pilot study is to assess the efficacy of minimally invasive autologous fat transfers at the amputation sites and the modulation of pain at the respective sites. Our investigators hypothesize that autologous fat grafting can provide a minimally invasive therapy to effectively mitigate pain syndromes at amputation sites, by introducing volume stable subcutaneous tissue over bony prominences and peripheral nerve trunks, thereby avoiding major surgical revisions and preserving limb length. The investigators further hypothesize that enriching the fat graft with autologous adipose stromal cells, a regenerative medicine approach, will lead to improved retention of the fat graft over time and result in a more favorable outcome.

The Investigators will evaluate:

1. Treatment of painful amputation sites in 5 patients with fat grafting, intended to provide additional subcutaneous tissue padding over bony structures and nerve trunks. Limb anatomy and healing of the graft over time, along with stability/persistence of the new tissue, will be assessed by high resolution CT scanning with 3D reconstruction. Patients will be followed for 24 months after treatment to define long term outcomes. Patients will be enrolled who have pain at an amputation site that limits function and/or interferes with the ability to use a prosthesis.
2. Biologic properties of the cells within the fat graft and correlate with clinical outcomes. This will include adipose stem cell yield per volume of fat tissue, cell proliferation, capacity for adipogenic differentiation, lipolysis, and cell sub-population analysis by multiparameter flow cytometry. Results of these assays will be correlated with graft volume retention to search for predictors of good clinical outcome that are related to variation on adipose biology between subjects.
3. Quality of life measurements in patients before and after autologous fat grafting using validated psychosocial measures. This will include SF 36, the Beck inventory, and instruments designed for assessing limb function.

DETAILED DESCRIPTION:
Traumatic amputations are prevalent and pose many challenges for our wounded warriors. A recent publication reported that during the current conflicts, over 950 military personnel have sustained combat-related amputations, with 15% of them occurring more than 12 weeks after initial injury (1). Updated statistics place this number of amputees at over 1050 (personal communication, COL Paul Pasquina, Chief of the Integrated Department of Orthopaedics and Rehabilitation, Walter Reed National Military Medical Center-WRNMMC). The ability of a wounded warrior to gain optimal function after an amputation most often depends on his or her ability to successfully fit and adapt to a prosthesis. Once out of the acute phase, many patients with amputations suffer from pain when wearing a prosthesis, either from thin soft tissue cover over bony structures or peripheral nerves not well padded with soft tissue. Extrinsic residual limb pain is usually mechanical in origin related to the prosthetic socket or other prosthetic components. It is often the result of a mismatch between residual limb tissue tolerance and the prosthetic loads on the soft tissues. This sensitivity is often accentuated by superficial nerve trunks or neuromas at severed nerves that are exposed to excessive external mechanical loading (2). Poor socket interface, secondary skin breakdown, and/or pain may severely limit function.

This presents a very difficult clinical problem and historically, when possible, the clinical procedure would be to involve the surgical revision of the amputation site with associated shortening of the bone, lengthy scars, and prolonged healing. If a below the knee amputation has to be converted to an above knee level, then there are serious functional implications. For local tissues at the amputation site that are of poor quality (e.g. scarred or covered with a skin graft), a distant muscle flap may be required (3,4). These flaps may require transfer to the amputation site using microvascular anastomosis of the blood vessels. The procedure is highly invasive and can add the morbidity of decreased function, deformity, and risk of wound healing problems at the muscle donor site. Failure rates in lower limb flaps can be as high as 18.5% (5, 6). Flap ulceration rates tend to be higher in these weight-bearing flaps, both skin and muscle free flaps frequently need secondary debulking procedures to improve function, and painful neuromas are not uncommon (6,7).

A clinical solution that allows for the minimally invasive generation of new soft tissue padding at an amputation site without the need for further limb shortening, lengthy scars, a prolonged recovery, and significant donor site morbidity would have the potential to significantly help our wounded warriors and change clinical practice.

Autologous fat grafting as a potential solution. Grafting of autologous fat tissue is a minimally invasive surgical technique that starts with the harvest of fat tissue from the abdomen or thighs using liposuction through incisions less than 5mm in length. The lipoaspirate is then processed to concentrate the adipose fraction and reinjected into the donor site. This surgical procedure involves the immediate transplantation of a patient's own tissue in a single operative procedure. It has the advantages of:

* Minimal access incisions
* Ability to transfer significant amounts of tissue (hundreds of grams of tissue)
* Can be used in setting of previous surgical procedures and presence of hardware
* Usually performed as outpatient procedure
* Minimal donor site morbidity at graft harvest site
* Low risk compared with more invasive surgical procedures
* Can be repeated multiple times, if necessary, even using the same donor sites

The transfer of autologous tissues is not a new concept but just another method as we have seen with many types of flaps using various combinations of muscle, fat and skin have been well documented. Tissue flaps come from many different locations, and are used in many different ways to accomplish the desired results. Flaps have their own blood supply, they are more resilient than skin grafts, and usually produce much better results from a cosmetic standpoint because they can provide a better match for skin tone and texture. Skin flaps are also a better choice when tissue "bulk" is needed to fill contour defects. The obvious advantage is to use autologus tissue versus xenografts and allografts; each having known risks of rejection and adverse events.

The literature has unequivocally demonstrated that clinical fat grafting in buttocks (a similar weight-bearing anatomic region) can be performed safely and effectively with retention rates approximating 75% up to 2 years and beyond (23-25). In an OVID database search of fat grafting articles, over 9000 articles have referenced the use of fat grafts in a wide arena of clinical situations. Specifically to this application over 100 references were relevant to this proposal and provided below.(26-132)

The investigators propose a clinical trial to assess the efficacy of minimally invasive autologous fat transfer for addressing pain and poor prosthetic fit at amputation sites. This surgical procedure involves the immediate transplantation of a subject's own tissue and does not require FDA oversight. Importantly, we will use our knowledge and expertise working with adipose stromal cells to compare a regenerative medicine cell therapy modification of the fat grafting procedure with more traditional fat graft preparations.

The biggest problem associated with fat grafting is unpredictable rates of fat graft resorption. This is likely related to the ability of the regenerating adipose tissue to rapidly develop a new blood supply. In this study, we will test a regenerative medicine approach of enriching the adipose graft with autologous adipose stem cells (stromal cell enriched adipose grafting). This may serve to improve graft retention over time and potentially improve functional outcomes.

A modified preparation of the fat graft involves concentrating the endogenous stromal cells in the graft material in an effort to increase graft retention over time. The aspirated fat material used for fat grafting consists of mature adipocytes, a small amount of fibrous tissue, and immature adipose stromal cells (ASCs). These adipose stromal cells are a mixed population of non-lipid laden cells that serve to turn over mature adipocytes and vascular elements. "Preadipocytes," as well as endothelial precursor cells and multilineage progenitor cells, are found. Of note, ASCs have been shown to stimulate angiogenesis when stressed under hypoxic conditions and these cells may be instrumental in healing and volume retention of fat grafts. Yoshimura, et. al. (133) found that fat aspirated with a liposuction cannula (i.e. the method of fat harvest for fat grafting) is deficient in ASCs compared to whole fat. This is due to the fact that a major portion of ASCs are located around larger blood vessels that are left intact in the donor site after liposuction with a blunt cannula. The relative lack of ASCs in lipoaspirate may explain problems with fat graft reabsorption over time. Enriching lipoaspirate with ASCs should increase angiogenesis and, therefore, fat graft retention. This cell therapy approach takes advantage of the innate ability of ASC's to both secrete angiogenic factors and also differentiate into mature adipocytes. The improved blood vessel ingrowth can result in improved graft volume retention and superior reconstructive outcomes.

Our group at the University of Pittsburgh has developed clinically useful and scalable GMP methods for ASC extraction under an NIH funded program, led by Dr. Rubin (Co-Director of the Adipose Stem Cell Center) in collaboration with Dr. Albert Donnenberg, director of the clinical laboratories for cell processing. We are currently starting a fully funded project with the Armed Forces of Regenerative Medicine (AFIRM). We are utilizing our extraction techniques to perform ASC enriched fat grafting for facial trauma reconstruction and this has received IRB approval at our institution. This process is regulated under human cells, tissues and cellular and tissue-based products (HCT/P) guidelines under section 361 of the CFR (21CFR1271.10). HCT/P therapies are exempt from the requirement for the submission of an Investigational New Drug (IND) application.

For this project proposal, we have expanded the team to encompass expertise in reconstructive fat grafting, lower extremity reconstruction, physical medicine and rehabilitation, prosthetic design, nutritional support, and evaluation of psychosocial outcomes. Given the initial success with autologous fat grafting for facial reconstruction after trauma (analysis ongoing), even without enrichment of the graft with adipose stromal cells, we believe this therapy can be effectively applied for the treatment of limb pain. This procedure can be performed on an outpatient basis with no significant incisions on the limb, only small port sites measuring less than 5 mm. It is noted that this is a completely new, experimental application of a conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and able to provide informed consent
2. Have suffered injury resulting in an amputation with pain that limits the fitting and use of a prosthesis, despite maximal attempts to refit the prosthesis and/or change the design of the prosthesis
3. Be at least 3 months post-injury or post-surgery (from trauma procedures) so that acute edema is resolved
4. Soft tissue deficiencies are noted at amputation stump and are covered by intact skin
5. Willing and able to comply with follow up examinations, including radiographic studies
6. Active military
7. Able to provide informed consent

Exclusion Criteria:

1. Age less than 18 years
2. Patient has inability to provide informed consent process.
3. Amputated limb area intended for treatment has open wounds, tunneling or drainage with active infection unresolved with one course of antibiotic treatment.
4. Active infection anywhere in the body
5. Diagnosed with cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment
6. Known coagulopathy symptoms /diagnosis
7. Systemic disease that would render the fat harvest and injection procedure, along with associated anesthesia, unsafe to the patient.
8. Pregnancy
9. History of Diabetes Mellitus
10. History of severe peripheral arterial disease
11. Diagnosis of Schizophrenia or Bipolar Disorder (Subjects who are found to be stable on medication and receive psychiatric clearance could be eligible for study participation per the Physician's discretion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-09-14 (Actual); Study Completion 2016-09-14 (Actual)

PRIMARY OUTCOMES:
Treatment of Painful Amputation Sites | 26 months
  1) Treat painful amputation sites in 5 patients with fat grafting, to provide additional subcutaneous tissue padding over bony structures and nerve trunks. Limb anatomy and healing of the graft over time, along with stability/persistence of the new tissue, will be assessed by high resolution CT scanning with 3D reconstruction. Patients will be followed for 24 months after treatment to define long term outcomes. Patients will be enrolled who have pain at an amputation site that limits function and/or interferes with the ability to use a prosthesis.

SECONDARY OUTCOMES:
Assessment of biological cell properties within fat graft | 20 years
  Assess biologic properties of cells within the fat graft and correlate with clinical outcomes to include adipose stem cell yield per volume of fat tissue, cell proliferation, capacity for adipogenic differentiation, lipolysis, and cell sub-population analysis by multiparameter flow cytometry. Assay results to be correlated with graft volume retention to search for predictors of good clinical outcome that are related to variation on adipose biology between subjects. Banked cells are stored for current assay or assay developed at a FUTURE date for correlation.
Quality of Life improvement | 26 months
  Measure quality of life in patients before and after autologous fat grafting using validated psychosocial measures. This will include SF 36, the Beck inventory, and instruments designed for assessing limb function.

CONTACTS AND LOCATIONS:
Overall Officials: J.Peter Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Kuntscher MV, Erdmann D, Homann HH, Steinau HU, Levin SL, Germann G. The concept of fillet flaps: classification, indications, and analysis of their clinical value. Plast Reconstr Surg. 2001 Sep 15;108(4):885-96. doi: 10.1097/00006534-200109150-00011. PMID 11547143
- [Background] Jensen TS, Krebs B, Nielsen J, Rasmussen P. Phantom limb, phantom pain and stump pain in amputees during the first 6 months following limb amputation. Pain. 1983 Nov;17(3):243-256. doi: 10.1016/0304-3959(83)90097-0. PMID 6657285
- [Background] Stinner DJ, Burns TC, Kirk KL, Scoville CR, Ficke JR, Hsu JR; Late Amputation Study Team. Prevalence of late amputations during the current conflicts in Afghanistan and Iraq. Mil Med. 2010 Dec;175(12):1027-9. doi: 10.7205/milmed-d-10-00102. PMID 21265314
- [Background] Perrot P, Bouffaut AL, Perret C, Connault J, Duteille F. Risk factors and therapeutic strategy after failure of free flap coverage for lower-limb defects. J Reconstr Microsurg. 2011 Mar;27(3):157-62. doi: 10.1055/s-0030-1268855. Epub 2010 Nov 23. PMID 21104612
- [Background] Weinberg MJ, Al-Qattan MM, Mahoney J. "Spare part" forearm free flaps harvested from the amputated limb for coverage of amputation stumps. J Hand Surg Br. 1997 Oct;22(5):615-9. doi: 10.1016/s0266-7681(97)80359-2. PMID 9752917
- [Background] Touam C, Rostoucher P, Bhatia A, Oberlin C. Comparative study of two series of distally based fasciocutaneous flaps for coverage of the lower one-fourth of the leg, the ankle, and the foot. Plast Reconstr Surg. 2001 Feb;107(2):383-92. doi: 10.1097/00006534-200102000-00013. PMID 11214053
- [Background] Goldberg JA, Adkins P, Tsai TM. Microvascular reconstruction of the foot: weight-bearing patterns, gait analysis, and long-term follow-up. Plast Reconstr Surg. 1993 Oct;92(5):904-11. PMID 8415972
- [Background] Coleman SR, Saboeiro AP. Fat grafting to the breast revisited: safety and efficacy. Plast Reconstr Surg. 2007 Mar;119(3):775-85; discussion 786-7. doi: 10.1097/01.prs.0000252001.59162.c9. PMID 17312477
- [Background] Spear SL, Wilson HB, Lockwood MD. Fat injection to correct contour deformities in the reconstructed breast. Plast Reconstr Surg. 2005 Oct;116(5):1300-5. doi: 10.1097/01.prs.0000181509.67319.cf. PMID 16217471
- [Background] Zheng DN, Li QF, Lei H, Zheng SW, Xie YZ, Xu QH, Yun X, Pu LL. Autologous fat grafting to the breast for cosmetic enhancement: experience in 66 patients with long-term follow up. J Plast Reconstr Aesthet Surg. 2008 Jul;61(7):792-8. doi: 10.1016/j.bjps.2007.08.036. Epub 2008 Mar 5. PMID 18321802
- [Background] Guyuron B, Majzoub RK. Facial augmentation with core fat graft: a preliminary report. Plast Reconstr Surg. 2007 Jul;120(1):295-302. doi: 10.1097/01.prs.0000264399.40701.71. PMID 17572578
- [Background] Hu S, Zhang H, Feng Y, Yang Y, Han X, Han X, Zhong Y, Shi J. Introduction of an easy technique for purification and injection of autogenous free fat parcels in correcting of facial contour deformities. Ann Plast Surg. 2007 Jun;58(6):602-7. doi: 10.1097/01.sap.0000248110.59452.49. PMID 17522480
- [Background] Kaufman MR, Bradley JP, Dickinson B, Heller JB, Wasson K, O'Hara C, Huang C, Gabbay J, Ghadjar K, Miller TA. Autologous fat transfer national consensus survey: trends in techniques for harvest, preparation, and application, and perception of short- and long-term results. Plast Reconstr Surg. 2007 Jan;119(1):323-331. doi: 10.1097/01.prs.0000244903.51440.8c. PMID 17255689
- [Background] Sardesai MG, Moore CC. Quantitative and qualitative dermal change with microfat grafting of facial scars. Otolaryngol Head Neck Surg. 2007 Dec;137(6):868-72. doi: 10.1016/j.otohns.2007.08.008. PMID 18036412
- [Derived] Bourne DA, Thomas RD, Bliley J, Haas G, Wyse A, Donnenberg A, Donnenberg VS, Chow I, Cooper R, Coleman S, Marra K, Pasquina PF, Rubin JP. Amputation-Site Soft-Tissue Restoration Using Adipose Stem Cell Therapy. Plast Reconstr Surg. 2018 Nov;142(5):1349-1352. doi: 10.1097/PRS.0000000000004889. PMID 30511990